CLINICAL TRIAL: NCT07234981
Title: PSMA-PET Guided De-escalation of Salvage Radiation Treatment in Patients With Recurrent Prostate Cancer After Prostatectomy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 733-25-FB
Record Dates: First submitted 2025-10-15; First posted 2025-11-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- De-escalated PSMA-guided salvage radiation (Experimental): Enrolled patients will receive an MRI and PSMA-PET/CT scan to identify locations of disease. The intervention will involve salvage radiation therapy to the prostate bed, pelvis, and pelvic nodes as indicated by imaging. External beam radiation therapy will consist of 45 Gy delivered in 25 daily fractions, followed by a sequential boost to PET-avid disease to 63-70.2 Gy in an additional 10-14 fractions.
  Interventions: Radiation: PSMA-guided Salvage Radiation

INTERVENTIONS:
Radiation: PSMA-guided Salvage Radiation — External beam radiation therapy will consist of 45 Gy delivered in 25 daily fractions, followed by a sequential boost to PET-avid disease to 63-70.2 Gy in an additional 10-14 fractions.

SUMMARY:
Purpose: Prospective, single-site Phase II study testing whether PSMA-PET/MRI-guided, de-escalated salvage radiation reduces acute Grade ≥2 toxicity versus a 44% historical rate, while maintaining cancer control after prostatectomy.Population/Eligibility: Adult men ≥30 years with prior radical prostatectomy and biochemical persistence/recurrence per NCCN (persistent positive PSA after RP, or undetectable PSA that becomes detectable and rises on ≥2 determinations, or PSA >0.1 ng/mL). Must have a targetable PSMA-avid lesion in the prostate bed and/or pelvic lymph nodes and/or an MRI-defined lesion suspicious for local recurrence. KPS ≥80 or ECOG ≤2; life expectancy >5 years; able to consent. Exclude: Evidence of distant metastatic disease outside pelvic nodes (including osseous involvement), conditions that preclude radiation, or factors preventing protocol compliance.Interventions & Evaluations: Baseline history/physical, vitals, performance status, labs (PSA, CBC w/diff, CMP/creatinine), pelvic MRI and PSMA-PET/CT; optional biopsy if feasible. External beam radiation therapy (LINAC/VMAT) with daily image guidance: pelvis 45 Gy in 25 fractions, followed by a sequential boost to PSMA/MRI-defined disease to 63-70.2 Gy in 10-14 additional fractions, with protocolized OAR constraints. All participants receive standard-of-care androgen deprivation therapy (ADT) for 6-24 months at the treating clinician's discretion. Weekly on-treatment visits; physician-assessed toxicities graded by CTCAE v5. Patient-reported outcomes (IPSS; FACT-P) at baseline and each in-person follow-up.Follow-up: Phone toxicity check 1 month post-RT; clinic at 4 months post-RT, then every 3 months thereafter until 24 months after completion of ADT. At each visit: H&P, CTCAE toxicity assessment, and PSA. If biochemical failure occurs, imaging (PSMA-PET/CT, CT and/or MRI) is obtained per standard of care to assess clinical progression.Endpoints/Design: Primary endpoint: acute (≤4 months post-RT) Grade ≥2 toxicity (all types). Secondary endpoints: 2-year biochemical progression-free survival; chronic toxicity and patient-reported outcomes from 4-24 months; 24-month local control, locoregional control, distant metastasis, and overall survival. Simon optimal two-stage design with interim analysis after the first 18 patients complete RT (stop if ≥8 have Grade ≥2 acute toxicity); total planned enrollment up to 54.

ELIGIBILITY:
Inclusion Criteria:

1. Prior biopsy proven prostate cancer for which they underwent a radical prostatectomy with curative intent.
2. Evidence of biochemical recurrence as defined by NCCN: Persistent positive PSA post-radical prostatectomy (RP) or an undetectable PSA after RP with a subsequent detectable PSA that increases on ≥2 determinations (PSA recurrence) or increases to PSA >0.1 ng/mL.
3. Targetable PSMA-avid lesion within the prostate bed, pelvic lymph nodes, or both and/or targetable lesion in prostate bed defined on MRI suspicious for local recurrence.
4. If lesions are amenable for biopsy this may be attempted, but biopsy proven recurrence/persistence is not required for trial enrollment.
5. Life expectancy greater than 5 years.
6. Karnofsky performance status ≥ 80 or Eastern Cooperative Oncology Group performance status ≤ 2 within 14 days prior to registration.
7. Age ≥ 30 years.
8. Patient must be able to provide study-specific informed consent prior to study entry.

Exclusion Criteria:

1. Evidence of distant metastatic disease outside the pelvic lymph nodes (including osseous pelvic disease).
2. Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse.
3. Relative or absolute contraindications to radiation therapy as determined by the treating physician. These include but are not limited to inflammatory bowel disease, connective tissue disorders (systemic lupus erythematosus, scleroderma, etc.), and genetic disorders that risk increased sensitivity to radiation therapy.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer Only-Males
Enrollment: 54 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2029-06-05 (Estimated); Study Completion 2029-06-05 (Estimated)

PRIMARY OUTCOMES:
Grade 2+ acute toxicity occurence | 4 months
  Determine the impact of de-escalated PSMA-guided salvage radiation on grade 2+ acute toxicity (i.e., <4 months) compared to historical controls.

SECONDARY OUTCOMES:
Occurrence of biochemical progression-free survival | 2-years
  Determine if 2-year biochemical progression-free survival with de-escalated PSMA-guided salvage radiation is comparable to historical post-salvage radiation treatment.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2-years
  Evaluate chronic toxicity from de-escalated PSMA-guided salvage radiation from 4 months to 2 years.
Overall Survival | 2-years
  Evaluate 24-month local control, locoregional control, distant metastasis, and overall survival.
Comparison of patient reported outcomes pre-, during follow-up, and post-study using the IPSS (International Prostate Symptom Score) | 2-Years
  The IPSS (International Prostate Symptom Score) will be summarized using descriptive statistics at each time point collected as n, mean, SD, median, minimum, and maximum. Changes over time will be displayed graphically. Generalized linear mixed models will be used to look for changes over time while accounting for within subject correlation using a random effect. Scores for each question are tallied, a higher score is indicative of worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baine, PhD/MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No